CLINICAL TRIAL: NCT07235878
Title: Effects of 12-week Magnesium Supplementation on Peri-menopause Symptoms, Cognition, Sleep and Psychological Wellbeing - a Randomised, Placebo-controlled Trial
Brief Title: 12-week Magnesium Supplementation on Peri-menopause Symptoms, Cognition, Sleep, and Psychological Well-being
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northumbria University (Other)
Collaborators: Vitabiotics (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 10251
Record Dates: First submitted 2025-09-17; First posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Perimenopause; Perimenopausal Women; Perimenopause, Climacteric Syndrome
Keywords: perimenopause; cognition; psychological wellbeing; sleep; magnesium; memory
MeSH Terms: interventions — Magnesium Hydroxide

STUDY DESIGN:
Intervention Model Description: Active vs. placebo
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo capsule consumed for 84 days
  Interventions: Other: Placebo
- 375mg magnesium hydroxide (Experimental): Magnesium hydroxide capsule consumed for 84 days
  Interventions: Dietary Supplement: Magnesium hydroxide 375mg

INTERVENTIONS:
Other: Placebo — 12 week placebo supplement of 2 capsules per day
  Arms: Placebo
Dietary Supplement: Magnesium hydroxide 375mg — 12 week supplementation of 2 capsules per day of Magnesium hydroxide
  Arms: 375mg magnesium hydroxide

SUMMARY:
Perimenopause is a transition phase into menopause, characterised by menopausal symptoms while menstrual periods are still occurring. Common symptoms of perimenopause include hot flushes, night sweats, mood swings, anxiety, sleep disturbances, fatigue, and cognitive difficulties. These symptoms can be both frequent and intense, with the potential to significantly deteriorate women's quality of life. Despite an increase in public discourse around menopause, there are still large gaps in knowledge. Previous literature has suggested a relationship between diet and menopause management. However, studies in this area are limited and women often rely on social media for advice on supplements to address menopause complaints. One supplement that has received a lot of attention with purported benefits for menopause is magnesium, primarily due to its links to energy and or/sleep, however no studies have explored psychological effects of magnesium supplementation in perimenopause.

The aim of this study is to explore the effects of 12-weeks magnesium supplementation on perimenopause symptoms, cognition, sleep, and psychological well-being.

DETAILED DESCRIPTION:
The term "perimenopause" describes a woman's life stage during which she undergoes changes due to hormone fluctuations but has not yet gone a full year without menstruation. It is a normal aspect of aging that typically affects women between the ages of 45 and 55, although some women may experience it sooner. While each person experiences symptoms differently, some common symptoms include irregular periods, hot flushes, night sweats, mood fluctuations, difficulty sleeping, decreased libido, vaginal dryness, memory and concentration problems. One widely recognised treatment for managing menopause symptoms is hormone replacement therapy (HRT). Although the benefits of HRT generally outweigh the risks, alternative options are needed for those with a history of breast cancer. Concerns surrounding risks have led many women to explore alternative approaches, including botanical and dietary supplements despite limited research on their efficacy and long-term effects. Women are increasingly turning to social media for advice on how to manage symptoms, and supplement manufacturers are beginning to target this audience with claims that they can reduce menopause symptoms. There is evidence of a link between nutrition and menopause, however research in this area is limited, especially in perimenopause. Magnesium is commonly promoted as a treatment for menopause symptoms, and there is some evidence that it improves sleep and overall well-being, but no research has looked into its effects in perimenopause. This study aims to examine the effects of 12-week magnesium hydroxide supplementation on cognition, sleep and psychological well-being in peri-menopausal women, with the results compared with those of a placebo.

ELIGIBILITY:
Inclusion Criteria:

* Self-assess as healthy
* Report experiencing troublesome peri-menopause symptoms in the past 6 months but not post-menopausal (defined as 12 months with no periods)

Exclusion Criteria:

* Post-menopausal
* Lactating, pregnant or seeking to become pregnant
* Nut Allergy
* Taken antidepressant/antianxiety medication or other medication with strong likelihood for effects on cognition or sleep in the past 6 months.
* Habitual magnesium supplementation (defined as more than 3 consecutive days or 4 days in total). Will be excluded unless washout for 1 month.
* Menopause symptoms have been medically induced.
* Receiving gender-affirming hormone therapy.

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Estimated)
Dates: Start 2025-11-17 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Numeric working memory task % accuracy | Conducted at baseline (pre-dose), at 6 weeks post-dose, and at 12 weeks post-dose.
  Cognitive function - working memory task. Measured as a percentage, with a higher score indicating better performance.
Numeric working memory task reaction time | Conducted at baseline (pre-dose), at 6 weeks post-dose, and at 12 weeks post-dose.
  Cognitive function - working memory task. Measured as reaction time (in milliseconds), with a lower score indicating better performance.
3-back task % accuracy | Conducted at baseline (pre-dose), at 6 weeks post-dose, and at 12 weeks post-dose.
  Cognitive function - working memory task. Measured as a percentage, with a higher score indicating better performance.
3-Back task reaction time | Conducted at baseline (pre-dose), at 6 weeks post-dose, and at 12 weeks post-dose.
  Cognitive function - working memory task. Measured as reaction time (in milliseconds), with a lower score indicating better performance.
Corsi blocks task score | Conducted at baseline (pre-dose), at 6 weeks post-dose, and at 12 weeks post-dose.
  Cognitive function - working memory task. Scored as level of difficulty reached (4 upwards), with a higher score indicating better performance.
Alphabetic working memory task % accuracy | Conducted at baseline (pre-dose), at 6 weeks post-dose, and at 12 weeks post-dose.
  Cognitive function - working memory task. Measured as a percentage, with a higher score indicating better performance.
Alphabetic working memory task reaction time | Conducted at baseline (pre-dose), at 6 weeks post-dose, and at 12 weeks post-dose.
  Cognitive function - working memory task. Measured as reaction time (in milliseconds), with a lower score indicating better performance.
Word recognition % accuracy | Conducted at baseline (pre-dose), at 6 weeks post-dose, and at 12 weeks post-dose.
  Cognitive function - episodic memory. Measured as a percentage, with a higher score indicating better performance.
Word recognition reaction time | Conducted at baseline (pre-dose), at 6 weeks post-dose, and at 12 weeks post-dose.
  Cognitive function - episodic memory task. Measured as reaction time (in milliseconds), with a lower score indicating better performance.
Picture recognition % accuracy | Conducted at baseline (pre-dose), at 6 weeks post-dose, and at 12 weeks post-dose.
  Cognitive function - episodic memory task. Measured as a percentage, with a higher score indicating better performance.
Picture recognition reaction time | Conducted at baseline (pre-dose), at 6 weeks post-dose, and at 12 weeks post-dose.
  Cognitive function - episodic memory task. Measured as reaction time (in milliseconds), with a lower score indicating better performance.

SECONDARY OUTCOMES:
The Menopause-Specific Quality of Life Questionnaire (Hilditch, 1996) | Conducted at baseline (pre-dose), at 6 weeks post-dose, and at 12 weeks post-dose.
  Assesses the effect of menopausal symptoms on quality of life in four domains: vasomotor, psychosocial, physical, and sexual; as well as providing a total score. The questionnaire has 29 items, each item is a symptom of menopause, the participants rate each symptom between 0 (not at all bothered) to 6 (bothered all the time.) The vasomotor symptoms include items such as 'hot flushes' and 'sweating'; psychological symptoms include 'accomplishing less than I used to' and 'poor memory'; physical symptoms include 'difficulty sleeping' and 'weight gain'; sexual symptoms include 'vaginal dryness' and 'avoiding intimacy'. A conversion score is created for each of the 4 domains: vasomotor; psychosocial; physical; sexual; as well as a total score. Each score ranges from 1 -8, with higher scores indicating greater problems.
Centre for Epidemiologic Studies Depression Scale (Radlof, 1997) | Conducted at baseline (pre-dose), at 6 weeks post-dose, and at 12 weeks post-dose.
  This is an established questionnaire used to measure symptoms associated with depression. The questionnaire has 20 items, including 'my sleep is restless', 'I felt depressed' and 'I felt lonely'. The participants rate the symptom on a scale between <1 day and 5 to 7 days, the 4 scale points are: Rarely or none of the time (less than 1 day); Some or a little of the time (1-2 days); Occasionally or a moderate amount of time (3-4 days); Most or all of the time (5-7 days). The possible range of scores is between 0 to 60, higher scores indicate more presence of symptomatology. The scoring of positive items is reversed.
The State-Trait Anxiety Inventory, TRAIT subscale (Spielberger, 1983) | Conducted at baseline (pre-dose), at 6 weeks post-dose, and at 12 weeks post-dose.
  The state-trait anxiety inventory will be used to measure anxiety levels, specifically trait anxiety. It consists of 20 items and the scale ranges from 1 to 4: 1 = almost never, 2 = sometimes, 3 = often and 4 = almost always. The nine positive items will be reversed for scoring, items 21, 23, 26, 27, 30, 33, 34, 36 and 39. The possible range of scores is 20 to 80, higher scores indicate higher levels of trait anxiety within the participant. Examples of items within the questionnaire include: 'I feel like a failure' and 'I feel secure'.
The Perceived Stress Scale (Cohen et al., 1983) | Conducted at baseline (pre-dose), at 6 weeks post-dose, and at 12 weeks post-dose.
  This established questionnaire will be used to measure the perception of stress. Each of the ten items are rated on a scale between 0 (never) to 4 (very often.) The five scale points are 0 = never, 1 = almost never, 2 = sometimes, 3 = fairly often, 4 = very often. The four positive items will be reversed for scoring, items 4, 5, 7 and 8. The questionnaire item examples include 'In the last month, how often have you been upset because of something that happened unexpectedly?' and 'In the last month, how often have you felt that you were unable to control the important things in your life?'. The possible range of scores is between 0 to 40, higher scores indicate high participant perceived stress.
Visual Analogue Mood Scales (VAMS) | Conducted at baseline (pre-dose), at 6 weeks post-dose, and at 12 weeks post-dose.
  This is a series of mood scales. Each scale is a line anchored at either side by an adjective describing a mood. Participants must click at a point on the scale that represents how they are feeling at that point in time. There are 18 scales in total, each scored out of 100. From these scales three composite scores are calculated describing feelings of 'Alertness', 'Stress' and 'Tranquillity', which are also presented as a score out of 100.
Sleep Related Impairment (PROMIS-SRI) (Yu et al., 2011) | Conducted at baseline (pre-dose), at 6 weeks post-dose, and at 12 weeks post-dose.
  The PROMIS-SRI will be used to measure sleep related impairment. The questionnaire contains 8 items, and participants are required to answer in relation to their sleep within the past 7 days. Each item is rated on a scale from 1-5. The items are then summed to create a single value (range 8-40), with higher scores indicating higher levels of sleep disturbance. Examples of items within the questionnaire include: 'I felt alert when I woke up' and 'I had a hard time getting things done because I was sleepy'.
Sleep Disturbance (PROMIS-SD) (Yu et al., 2011) | Conducted at baseline (pre-dose), at 6 weeks post-dose, and at 12 weeks post-dose.
  The PROMIS-SD will be used to measure sleep disturbance. The questionnaire contains 8 items, and participants are required to answer in relation to their sleep within the past 7 days. Each item is rated on a scale from 1-5. The items are then summed to create a single value (range 8-40), with higher scores indicating higher levels of sleep disturbance. Examples of items within the questionnaire include: 'my sleep was restless' and 'I had difficulty falling asleep'.

CONTACTS AND LOCATIONS:
Locations (1):
- School of Psychology, Northumbria University, Newcastle upon Tyne, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
An anonymised dataset will be shared on this platform within the results section. Any information which may identify individual participants will be removed from the dataset before it is shared. Data will be shared in accordance with FAIR (findable, accessible, interoperable, reusable) principles. Participants will consent to the data being shared in this way.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available 3 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis.
Access Criteria: Fully accessible